CLINICAL TRIAL: NCT01250938
Title: 2/2-Effects of Parent-Implemented Intervention for Toddlers With Autism Spectrum
Brief Title: Effectiveness of Early Intervention in an Underserved Population
Acronym: ESI-CO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Autism Speaks (Other); Florida State University (Other)
Responsible Party: Principal Investigator, Catherine Lord, Ph.D., Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1108011843; Autism Speaks 5766 (Other Grant/Funding Number: Autism Speaks); R01MH078165 (NIH)
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorders
Keywords: autism; autism spectrum disorders; pervasive developmental disorders; intervention; low-income; underserved populations; underrepresented populations
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Child Development Disorders, Pervasive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ESI - Community Outreach (Experimental): All families receive the same Early Social Intervention - Community Outreach (ESI-CO) treatment for 3 months in addition to 6 months of community resource support.
  Interventions: Behavioral: ESI - Community Outreach

INTERVENTIONS:
Behavioral: ESI - Community Outreach — This is an individualized caregiver-implemented intervention (ESI-CO) offered in 2 weekly sessions to teach caregivers how to embed strategies to support social communication skills within everyday routines, activities, and places for 3 months. Additionally, families receive 6 months (3 months during weekly home sessions and three months upon the completion of weekly home sessions) of resource support to identify local and community autism programs available for continued intervention and services.
  Other Names: Modified ESI

SUMMARY:
The purpose of this study is to test the applicability of a caregiver-implemented autism intervention protocol to a deliberately recruited low-income, underserved population.

DETAILED DESCRIPTION:
Families of racial/ethnic minority, lower levels of education, and those who live in non-metropolitan areas have been found to experience greater limitations in accessing services for Autism Spectrum Disorder (ASD) (Thomas, Ellis, McLaurin, Daniels, & Morrissey, 2007). Black and Hispanic children have been found to have lower odds of having a documented ASD classification than white children (Mandell, Wiggins, Arnstein Carpenter, Daniels, Durkin et al., 2009) and of those children who do receive an ASD diagnosis, many of them are not diagnosed in early childhood. The age of first ASD diagnosis received has been found to be significantly higher for African American and Latino children compared to white children (Mandell, Listerud, Levy, & Pinto-Martin, 2002). For these reasons, it is important that the effectiveness of intensive early intervention for children with ASD is examined across varying cultural and socioeconomic backgrounds.

This project is directed by Dr. Catherine Lord at the University of Michigan, in collaboration with Dr. Amy Wetherby at Florida State University to test the applicability of a modified caregiver-implemented autism intervention (Modified Early Social Interaction; ESI) to a deliberately recruited low-income, underserved population. UM will recruit 28 children and FSU will recruit 16 children diagnosed with ASD who are between 24 and 42 months of age over a period of 3 years, totaling 44 caregiver-child dyads. This study will utilize a multiple baseline single-subject research design. Dyads will complete 1 month of weekly 1-hour baseline observations followed by three months of the modified ESI intervention. Child and family characteristics predicting response to intervention will be identified and findings will contribute to the development of autism interventions serving families from diverse backgrounds.

ELIGIBILITY:
Inclusion Criteria:

* caregiver(s) with less than a 4-year college degree
* family income equal to or below 2x the federal poverty line
* English as the predominantly-spoken language.
* child received diagnosis of autism spectrum disorder before treatment
* child is between 24 and 42 months at the start of treatment
* child has normal hearing and adequate motor control to make simple actions (giving, reaching)
* family agrees to 2-4 weeks of weekly 1-hour observations, 3 months of 2 intervention sessions per week, and 3 months of 1 intervention session per month.
* family agrees to pre-treatment, post-treatment, and follow-up evaluation and videotaping of intervention sessions and weekly video check during the treatment.

Exclusion Criteria:

-Must meet eligibility requirements stated above.

Ages: 24 Months to 54 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2009-07; Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Caregiver Transactional Support | Weekly
  Measures caregiver's development of behavioral strategies to support child's social and communicative behavior.

SECONDARY OUTCOMES:
Child Outcome | All measures pre-treatment, post-treatment, and at 3 month follow-up. Some measures weekly and monthly
  Child measures of autism symptoms, social communication, developmental level, and adaptive behavior.
Caregiver Outcome | All measures pre-treatment, post-treatment, and at 3 month follow-up. Some measures weekly and monthly
  Caregiver measures self-reported family functioning, resources, well-being and treatment adherence, fidelity, and satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Lord, Ph.D., Principal Investigator — Weill Medical College of Cornell University; Amy Wetherby, Ph.D., Principal Investigator — Florida State University
Locations (2):
- United States (2):
  - Florida State University, Tallahassee, Florida
  - Weill Cornell Medical College, White Plains, New York

IPD SHARING:
Plan to Share IPD: Yes
Data are maintained by Florida Statue University, the data coordinating center for this collaborative project. We have shared deidentified study data by depositing it in the NIH National Database for Autism Research (NDAR).
  We have a long-standing commitment to making our data available to other investigators. As part of our previous work with NIMH (e.g. NIMH Collaborative RO1 MH089390) and others (e.g. Simons Simplex Collection), our data collection methods and data structures have been designed with NDAR's data-sharing protocol in mind (we collect information necessary to generate the Global Unique Identifier). Our study uses standardized assessments and all data are maintained in a secure database.